CLINICAL TRIAL: NCT02312167
Title: Essai de faisabilité Pour Une Endomicroscopie Robotisée Dans la redéfinition Des Stratégies d&Apos;ExérèsE
Brief Title: Feasibility Study for Robotic Endomicroscopy to Better Define Resection Strategies (PERSEE)
Acronym: PERSEE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Mutualiste Montsouris (Other)
Collaborators: Mauna Kea Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MKT-2013-PERSEE-01
Record Dates: First submitted 2014-11-28; First posted 2014-12-09 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2014-12

CONDITIONS: Cancer of Digestive System; Ovarian Cancer
Keywords: endomicroscopy; optical biopsy; exploratory surgery; resection surgery; robot-assisted; peritoneum carcinosis; inflammatory; rectum cancer; liver cancer; ovarian cancer; digestive cancer; pancreas cancer; duodenum cancer
MeSH Terms: conditions — Digestive System Neoplasms; Ovarian Neoplasms; Rectal Neoplasms; Liver Neoplasms; Gastrointestinal Neoplasms; Pancreatic Neoplasms; Duodenal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- confocal laser endomicroscopy (Experimental): confocal laser endomicroscopy : 10 to 15 minutes endomicroscopy procedure to obtain real time microscopical images of healthy and malignant tissue of the targeted organs
  Interventions: Device: confocal laser endomicroscopy

INTERVENTIONS:
Device: confocal laser endomicroscopy — probe-based and needle-based confocal laser endomicroscopy
  Other Names: optical biopsy; Cellvizio

SUMMARY:
This study aims at demonstrating the feasibility of probe-based confocal laser endomicroscopy (pCLE) and needle-based confocal laser endomicroscopy (nCLE).

Contraindications for resection surgery may sometimes be missed during exploratory surgical procedures. That may lead to an incomplete thus useless surgery and delay the right treatment.

The objectives of this study are to improve the detection of cancer extension during exploratory procedures and to guide resection to ensure clear margins.

DETAILED DESCRIPTION:
This study involves several innovations including :

* the robotization of the confocal miniprobe for a better an d more precise handling of the probe
* the use of different contrast agent and administration mode (Fluorescein, Patented Blue V, Indocyanine Green via intravenous, interstitial or topical administration)
* the communication between the operative room and the pathologist room for a real time assessment by the surgeon and by the pathologist of the endomicroscopic images

ELIGIBILITY:
Inclusion Criteria:

* patient scheduled for an exploratory surgery or a resection surgery for an abdomino-pelvic cancer
* patient able to give written informed consent

Exclusion Criteria:

* allergy to fluorescein
* allergy to patented blue
* allergy to ICG
* previous life-threatening allergic reactions and known hypersensitivity
* pregnancy or breast-feeding
* history of cardio-pulmonary disease (including bronchial asthma)
* restricted renal function
* patient under a beta-blockers treatment
* patient who cannot give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
The number of participants with adverse events, their type and severity | 8 months

SECONDARY OUTCOMES:
The ease of manipulation of the robotized probe (grade 1 to 5) | 8 months
  during or after each procedure, the surgeon is asked to assess the ease of manipulation of the device

OTHER OUTCOMES:
the quality of real time communication between the pathologist lab and the OR (grade 1 to 5) | 8 months
  during or after each procedure, the surgeon and the pathologists are asked to assess the quality of audiovisual communication
number of interpretable images per organ, per contrast agent and per pathology | 8 months
  each sequence acquired during the cases will be annotated as to which organ it is, and the final diagnosis of the specimen (healthy, cancerous, inflammation, etc ...). Thanks to this, a more complete atlas of images obtained in digestive organs and conditions will be developed. This atlas will be used to describe image interpretation criteria for endomicroscopic images of various organs and conditions. This work will be done in conjunction by the investigators, the histopathologist, and an Mauna Kea Technologies representative familiar with image interpretation in current endomicroscopy indications.

CONTACTS AND LOCATIONS:
Overall Officials: Brice GAYET, MD, Principal Investigator — Mutualiste Montsouris Institute
Locations (1):
- Mutualiste Montsouris Institute, Paris, Paris, France

REFERENCES:
- [Derived] Fuks D, Pierangelo A, Validire P, Lefevre M, Benali A, Trebuchet G, Criton A, Gayet B. Intraoperative confocal laser endomicroscopy for real-time in vivo tissue characterization during surgical procedures. Surg Endosc. 2019 May;33(5):1544-1552. doi: 10.1007/s00464-018-6442-3. Epub 2018 Sep 19. PMID 30232616